CLINICAL TRIAL: NCT00681863
Title: Open Label Extension Study With Pramipexole (PPX) in Children With Tourette Syndrome
Brief Title: Open-label Extension Study of Pramipexole in the Treatment of Children and Adolescents With Tourette Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated for slow enrollment.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 248.642; 2008-000342-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Pramipexole; BID protein, human

ARMS (5):
- pramipexole 0.0625 mg BID (twice daily) (Active Comparator): all patients to receive one tablet of pramipexole 0.0625 mg BID for first 4 weeks (flexible dosing for all other arms)
  Interventions: Drug: pramipexole 0.0625 mg BID
- pramipexole 0.0625 mg QD (once daily) (Active Comparator): patients to receive one tablet of pramipexole 0.0625 mg QD
  Interventions: Drug: pramipexole 0.0625 mg QD
- pramipexole 0.125 mg BID (Active Comparator): patients to receive one tablet of pramipexole 0.125 mg BID
  Interventions: Drug: pramipexole 0.125 mg BID
- pramipexole 0.125 mg TID (three times daily) (Active Comparator): patients to receive one tablet of pramipexole 0.125 mg TID
  Interventions: Drug: pramipexole 0.125 mg TID
- pramipexole 0.25 mg BID (Active Comparator): patients to receive one tablet of pramipexole 0.25 mg BID
  Interventions: Drug: pramipexole 0.25 mg BID

INTERVENTIONS:
Drug: pramipexole 0.125 mg BID — titrated dose for those patients whose symptoms were not controlled on the 0.0625 mg BID dose
  Arms: pramipexole 0.125 mg BID
Drug: pramipexole 0.0625 mg QD — dose down titrated for those patients unable to tolerate the 0.0625 mg BID dosing
  Arms: pramipexole 0.0625 mg QD (once daily)
Drug: pramipexole 0.125 mg TID — titrated up for those patients whose symptoms were not adequately controlled on 0.125 mg BID dose
  Arms: pramipexole 0.125 mg TID (three times daily)
Drug: pramipexole 0.25 mg BID — titrated for those patients whose symptoms were not adequately controlled on 0.125 mg TID dose
  Arms: pramipexole 0.25 mg BID
Drug: pramipexole 0.0625 mg BID — 0.0625 mg BID given for first 4 wks of treatment
  Arms: pramipexole 0.0625 mg BID (twice daily)

SUMMARY:
The primary objective of this open-label, flexible dose study is to assess the safety and efficacy of pramipexole over a 24-week period in children and adolescents (age 6-17 years inclusive) diagnosed with Tourette Syndrome according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria and who have completed either Study 248.641 (NCT 00681863) or 248.644 (NCT 00558467).

ELIGIBILITY:
Inclusion criteria

1. Male or female patients aged 6-17 years at the time of enrollment into study 248.641 or 248.644 and who have completed study 248.641 or 248.644.
2. Written informed consent provided by the patient's parent (or legal guardian) and assent provided by the patient consistent with International Conference on Harmonization (ICH) Good Clinical Practice (GCP) and local Institutional Review Board (IRB) requirements for children obtained prior to any study procedures being performed.
3. Ability and willingness to comply with study treatment regimen and to complete study assessments.
4. Females of childbearing potential having a negative serum pregnancy test at Visit 1.
5. Females of childbearing potential must be using a medically accepted contraceptive method throughout the study. Acceptable methods of birth control are limited to: Intra-Uterine Device (IUD), oral, implantable, injectable contraceptives or estrogen patch, double barrier method (spermicide + diaphragm), or abstinence at the discretion of the investigator

Exclusion criteria

1. Breastfeeding females.
2. Development of any clinical condition in the preceding trial that in the investigator's opinion could be worsened by treatment with pramipexole.
3. Clinically significant renal disease or serum creatinine out of this range: 0.3 1.0 mg/dL for patients aged 3-12 years and 0.5-1.4 mg/dL for patients aged 13+ years.
4. Any of the following lab results at screening:

   Hemoglobin (Hgb) below lower limit of normal (LLN) which is determined to be clinically significant Basal thyroid stimulating hormone (TSH), triiodothyronine (T3) or thyroxine (T4) clinically significant (at the investigator's discretion) out of normal range at screening (if not caused by substitution therapy according the investigator's opinion) Patients with any clinically significant abnormalities in laboratory parameters at screening at the investigator's discretion.
5. Other clinically significant metabolic-endocrine, hematological, gastrointestinal disease, or pulmonary disease (such as severe asthma) in the opinion of the investigator that would preclude the patient from participating in this study.
6. History or presence of schizophrenia or any psychotic disorder. History or presence of any psychiatric disorder requiring medical therapy with the exception for patients with a diagnosis of Tourette Syndrome (TS), Attention Deficit Hyperactivity Disorder (ADHD) or Obsessive Compulsive Disorder (OCD) who are not on therapy other than pramipexole.
7. History or presence of clinical signs of epilepsy or seizures other than fever-related seizures in early childhood.
8. History or presence of clinical signs of any malignant neoplasm including suspicious undiagnosed skin lesion (which may be melanoma), melanoma, or a history of melanoma.
9. History of any other medical treatment for TS besides the study medication within 28 days prior to the baseline visit (14 days prior to baseline for guanfacine, 14 days prior to baseline for dopamine agonists, 14 days prior to baseline for L-Dopa, 35 days prior to baseline for fluoxetine).
10. Patients receiving psychotherapy are excluded unless they started the treatment at least 3 months prior to starting the trial and no changes in treatment are planned for the duration of the study.
11. Allergic response to pramipexole or the inactive ingredients in its tablet formulation.
12. Non-compliance with study medication (defined as less than 80% or more than 120%) during the preceding Study 248.641 or 248.644.
13. Concurrent participation in another clinical trial using any investigational drug since completion of the preceding Study 248.641 or 248.644.
14. Any other conditions, that in the opinion of the investigator, would interfere with the evaluation of the results or constitute a health hazard for the patient.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (14):
- United States (13):
  - 248.642.0026 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 248.642.0025 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 248.642.0006 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 248.642.0005 Boehringer Ingelheim Investigational Site, Cambridge, Massachusetts
  - 248.642.0003 Boehringer Ingelheim Investigational Site, Manhasset, New York
  - 248.642.0009 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.642.0018 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.642.0013 Boehringer Ingelheim Investigational Site, Orangeburg, New York
  - 248.642.0029 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 248.642.0010 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 248.642.0030 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 248.642.0008 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 248.642.0023 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
- 248.642.49004 Boehringer Ingelheim Investigational Site, Ulm, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole: 4 weeks individual dose titration starting with 0.0625 mg BID (twice daily), down-titration to 0.0625 QD (once daily) if not tolerated, and next steps 0.125 mg BID, 0.125 mg TID (three times daily) and 0.25 mg BID, according to efficacy assessment; established optimal dose for the remainder of the 24-week treatment period.
Period: Overall Study
Arm/Group | Pramipexole
Started | 45
Completed | 22
Not Completed | 23
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 2
Not completed — Other | 18

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) included all patients who were entered, were dispensed study medication and were documented to have taken at least one dose of study medication.
Groups:
- Pramipexole: 4 weeks individual dose titration starting with 0.0625 mg BID, down-titration to 0.0625 QD if not tolerated, and next steps 0.125 mg BID, 0.125 mg TID and 0.25 mg BID, according to efficacy assessment; established optimal dose for the remainder of the 24-week treatment period.
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.8 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5
  White | 40
Duration of Tourettes Syndrome [Number; unit: Participants]
  More than 5 years | 10
  Less than 1 year | 15
  1 to 5 years | 20
Height [Mean (Standard Deviation); unit: centimeters] | 152.6 (19.4)
Weight [Mean (Standard Deviation); unit: kilograms] | 53.01 (21.58)
Body mass index [Mean (Standard Deviation); unit: kilograms/square meter] | 22.064 (5.930)
Body temperature [Mean (Standard Deviation); unit: Degrees centigrade] | 36.752 (0.718)
Respiration [Mean (Standard Deviation); unit: breaths/minute] | 17.4 (2.0)
Obsessive Compulsive Disorder [Number; unit: Participants] — Diagnosis of disorder was performed using National Institute of Mental Health Diagnostic Interview Schedule for Children (NIMH DISC-IV)
  Participants
    Positive | 4
    Intermediate | 4
    Negative | 37
Attention Deficit Hyperactive Disorder [Number; unit: participants] — Diagnosis of disorder was performed using National Institute of Mental Health Diagnostic Interview Schedule for Children (NIMH DISC-IV)
  participants
    Positive | 17
    Intermediate | 6
    Negative | 22
Treatment received in previous trial (NCT00558467) [Number; unit: Participants]
  Received placebo | 14
  Received pramipexole | 31

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: Total Tic Score is the sum of ten individual ratings of the impairment due to tics. Each scale ranges from 0 (None/Absent) to 5 (Severe) and total score ranges from 0 to 50.
Time Frame: baseline and week 24
Population: The Full Analysis Set (FAS) with last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
Score on a scale | -9.8 (8.9)

2. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: Total Score is a rating of the overall impairment due to motor and phonic tics. The scale ranges from 0 (None) to 50 (Severe).
Time Frame: baseline and Week 24 (end of treatment visit)
Population: The Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
Score on a scale | -22.0 (21.0)

3. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and Week 1
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
Score on a scale | -7.2 (8.5)

4. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and Week 2
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
Score on a scale | -8.3 (7.7)

5. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and Week 3
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 44
Score on a scale | -8.6 (8.6)

6. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and week 4
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 44
Score on a scale | -9.3 (9.7)

7. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and Week 8
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 41
Score on a scale | -10.7 (9.4)

8. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and Week 12
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 35
Score on a scale | -12.3 (9.0)

9. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and Week 16
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 32
Score on a scale | -12.4 (9.3)

10. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and Week 20
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 26
Score on a scale | -11.7 (11.3)

11. Secondary Outcome: Mean Change From Baseline in Total Tic Score (TTS) of the Yale Global Tic Severity Scale
Description: as for outcome 1
Time Frame: baseline and Week 24
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
Score on a scale | -9.3 (10.4)

12. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 1
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
Score on a scale | -14.5 (18.2)

13. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 2
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
Score on a scale | -17.4 (17.6)

14. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 3
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 44
Score on a scale | -18.4 (19.8)

15. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 4
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 44
Score on a scale | -20.9 (21.5)

16. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 8
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 41
Score on a scale | -22.4 (21.9)

17. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 12
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 35
Score on a scale | -27.7 (20.9)

18. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 16
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 32
Score on a scale | -28.3 (20.2)

19. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 20
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 26
Score on a scale | -26.7 (24.9)

20. Secondary Outcome: Mean Change From Baseline in Total Score of the Yale Global Tic Severity Scale
Description: as for outcome 2
Time Frame: baseline and Week 24
Population: Observed Cases Full Analysis Set (OC FAS). All participants in FAS having observed data at the particular timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 22
Score on a scale | -22.0 (23.6)

21. Secondary Outcome: Clinical Global Impressions - Severity of Illness
Description: Overall improvement during the last week compared to baseline ranging from 1 (very much improved), 2 (much improved), to 7 (very much worse). Responder has 'very much' or 'much' improvement. Non responder has less improvement than 'much' improvement.
Time Frame: week 24
Population: The Full Analysis Set (FAS) with last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 42
score on a scale | -1.1 (1.1)

22. Secondary Outcome: Clinical Global Impressions - Severity of Illness, Categorized
Description: Assessment of the overall severity of illness on a scale ranging from 1 (not at all ill) to 7 (among the most extremely ill patients).
  Overall improvement during the last week compared to baseline ranging from 1 (very much improved), 2 (much improved), to 7 (very much worse). Responder has 'very much' or 'much' improvement. Non responder has less improvement than 'much' improvement.
Time Frame: week 24
Population: The Full Analysis Set (FAS) with last observation carried forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 42
participants
  Improved (change score <= -2) | 11
  Unchanged (change score of -1, 0, or +1) | 31
  Worsened (change score >= +2) | 0

23. Secondary Outcome: Clinical Global Impressions - Improvement
Description: Assessment of the overall improvement during the last week compared to the patient's condition at baseline on a scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: week 1
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

24. Secondary Outcome: Clinical Global Impressions - Improvement
Description: as for outcome 23
Time Frame: week 2
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

25. Primary Outcome: Patients With Adverse Events Leading to Discontinuation of Trial Drug
Description: Number of patients with Adverse Events leading to discontinuation of trial drug
Time Frame: 24 Weeks
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
participants | 1

26. Secondary Outcome: Clinical Global Impressions - Improvement
Description: as for outcome 23
Time Frame: week 3
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

27. Secondary Outcome: Clinical Global Impressions - Improvement
Description: as for outcome 23
Time Frame: week 4
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

28. Secondary Outcome: Clinical Global Impressions - Improvement
Description: as for outcome 23
Time Frame: week 8
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

29. Secondary Outcome: Clinical Global Impressions - Improvement
Description: as for outcome 23
Time Frame: week 12
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

30. Secondary Outcome: Clinical Global Impressions - Improvement
Description: as for outcome 23
Time Frame: week 16
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

31. Secondary Outcome: Clinical Global Impressions - Improvement
Description: as for outcome 23
Time Frame: week 20
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

32. Secondary Outcome: Clinical Global Impressions - Improvement
Description: as for outcome 23
Time Frame: week 24
Population: The Full Analysis Set (FAS) with last observation carried forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
participants
  Responder (Much improved or Very much improved) | 22
  Not Responder | 23

33. Secondary Outcome: Patient Global Impression - Improvement
Description: Assessment of the change of the patient's overall condition during the last week compared to the patient's condition at baseline on a scale ranging from 1 (very much better) to 7 (very much worse). A responder is defined as having a response of very much (1) or much better (2).
Time Frame: week 1
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

34. Secondary Outcome: Patient Global Impression - Improvement
Description: as for outcome 33
Time Frame: week 2
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

35. Secondary Outcome: Patient Global Impression - Improvement
Description: as for outcome 33
Time Frame: week 3
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

36. Secondary Outcome: Patient Global Impression - Improvement
Description: as for outcome 33
Time Frame: week 4
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

37. Secondary Outcome: Patient Global Impression - Improvement
Description: as for outcome 33
Time Frame: week 8
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

38. Secondary Outcome: Patient Global Impression - Improvement
Description: as for outcome 33
Time Frame: week 12
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

39. Secondary Outcome: Patient Global Impression - Improvement
Description: as for outcome 33
Time Frame: week 16
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

40. Secondary Outcome: Patient Global Impression - Improvement
Description: as for outcome 33
Time Frame: week 20
Population: This outcome measure was not analyzed due to the premature ending of the trial.
Arm/Group | Pramipexole
Number analyzed (Participants) | 0

41. Secondary Outcome: Patient Global Impression - Improvement
Description: as for outcome 33
Time Frame: week 24
Population: The Full Analysis Set (FAS) with last observation carried forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 45
participants
  Responder (Much better or Very much better) | 17
  Not Responder | 28

42. Secondary Outcome: Frequency of Patients With Possible Clinically Significant Abnormalities for Laboratory Parameters
Description: Frequency of patients with possible clinically significant abnormalities for laboratory parameters (blood hematology and electrolyte assessments, serum chemistry, including follicle-stimulating hormone (FSH), luteinizing hormone (LH) and estradiol for pubertal female patients, prolactin in all patients, testosterone in pubertal male patients, urine analysis)
Time Frame: Baseline and 24 weeks
Population: Observed Cases Treated set (OC TS). All participants in Treated Set having observed data at the particular timepoint.
Measure: Number; unit: participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 43
participants
  Haemoglobin - decrease | 2
  Eosinophils - increase | 3
  Phosphate - increase | 2
  Alkaline phosphatase - increase | 1

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Description: At each visit, the Investigator asked the patient and parent(s) (legal guardians) to elucidate any adverse events that may have occurred since the last visit in order to document if any adverse events had occurred, and carefully recorded the adverse event information reported.
Arm/Group | Pramipexole
Serious Adverse Events (participants affected / at risk) | 1/45
Other Adverse Events (participants affected / at risk) | 35/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=45)
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=45)
Abdominal pain upper (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 6
Pyrexia (General disorders) | 4
Hypersensitivity (Immune system disorders) | 4
Nasopharyngitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 4
Skin laceration (Injury, poisoning and procedural complications) | 3
Increased appetite (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 9
Somnolence (Nervous system disorders) | 3
Tic (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Orthostatic hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
The sponsor cancelled this trial prematurely. Thus, enrollment for 248.642 (NCT00681863) was significantly less than what was planned (120 planned vs. 45 entered). Therefore, the objectives of this study could not be fully assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract